CLINICAL TRIAL: NCT03867604
Title: Ultrasound-guided Fascial Release Injection for Myofascial Pain Syndrome in the Upper Trapezius Muscle: A Pilot Study
Brief Title: Ultrasound-guided Fascial Release Injection for Myofascial Pain Syndrome in the Upper Trapezius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N201811013
Record Dates: First submitted 2019-01-21; First posted 2019-03-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2019-01

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham injection (Sham Comparator): Subcutaneous injection at upper trapezium muscle level
  Interventions: Procedure: Sham injection
- Fascia injection (Experimental): Fascia injection, below upper trapezium muscle
  Interventions: Procedure: Fascia injection

INTERVENTIONS:
Procedure: Sham injection — Injection to the subcutaneous layer at upper trapezium level
  Arms: Sham injection
Procedure: Fascia injection — Injection to the fascia below upper trapezium muscle
  Arms: Fascia injection

SUMMARY:
Patients with myofascial pain syndrome at upper trapezius will be randomized into 2 groups, fascial injection group and subcutaneous control injection group. Pain condition pain, range of motion and function will be evaluated in 1 week, 4 weeks and 12 weeks after injection.

DETAILED DESCRIPTION:
Myofascial pain syndrome(MPS) is characterized by a trigger point with a hyperirritable nodule and taut band of muscle or fascia. MPS was usually treated by dry needling or met needing, local anesthetics injection, to the trigger point. According to recent researches, dry and wet needling to affected muscle are effectiveness for short term and medium term pain relief. Although some researches indicated an increased viscosity at fascial layer in MPS and there are few studies of manipulation for fascial release. There is not study of injective fascial release.

Investigators will include 40 patients with myofascial pain syndrome at upper trapezius. Participants will be randomized into 2 groups, fascia injection group and subcutaneous control injection group. Investigators will use algometer to measure pain threshold and peak pressure, measure the range of motion of neck and shoulder and assess the neck and shoulder function by questionnaire. The examination will be done before injection, immediately after injection, 1 week, 4 weeks and 12 weeks after injection.

To our hypothesis, investigators suggest focal anesthetics injection could decrease the fascial viscosity and improved pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years old
* diagnosed as a myofascial pain syndrome at upper trapezium muscle
* trigger point
* taut band
* refer pain while taut band irritation

Exclusion Criteria:

* Cognitive impairment.
* Post operation at neck and shoulder.
* Nerve compression at cervical region.
* Could not receive injection therapy, history of fainting during needling

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Upper back or shoulder pain | Change from baseline VAS at 1 week
  visual analogue scale(VAS), range 0-10, the higher the worse pain
Upper back or shoulder pain | Change from baseline VAS at 4 week
  visual analogue scale(VAS), range 0-10, the higher the worse pain
Upper back or shoulder pain | Change from baseline VAS at 12 week
  visual analogue scale(VAS), range 0-10, the higher the worse pain

SECONDARY OUTCOMES:
Function | Change from baseline SPADI at 1 week
  Shoulder Pain and Disability Index (SPADI), range 0-130, the higher the worse
Function | Change from baseline SPADI at 4 week
  Shoulder Pain and Disability Index (SPADI), range 0-130, the higher the worse
Function | Change from baseline SPADI at 12 week
  Shoulder Pain and Disability Index (SPADI), range 0-130, the higher the worse

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Cheng, Cheng, Study Director — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei medical university, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hsu CY, Hsu T, Lin YN, Cheng YH. Additional Effect of Interfascial Hydrodissection With Dextrose on Shoulder and Neck Function in Patients With Myofascial Pain Syndrome: A Randomized Control Trial. Am J Phys Med Rehabil. 2024 Sep 1;103(9):827-834. doi: 10.1097/PHM.0000000000002442. Epub 2024 Jan 31. PMID 38320240